CLINICAL TRIAL: NCT04592640
Title: Effects of Human Amniotic Mesenchymal Stem Cells (hAMSCs) on Wound Healing in Uremic Calciphylaxis Patients: an Open Label Single Arm Study
Brief Title: Stem Cells for Uremic Calciphylaxis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ningning Wang (Other)
Responsible Party: Sponsor-Investigator, Ningning Wang, Professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Stem cell
Record Dates: First submitted 2020-10-03; First posted 2020-10-19 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases; Calciphylaxis; Calcific Uremic Arteriolopathy; Treatment
Keywords: Chronic Kidney Diseases; Calciphylaxis; Calcific Uremic Arteriolopathy; Human Amniotic Mesenchymal Stem Cells; Rare disease (ORPHA280062)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Calciphylaxis; Rare Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uremic Calciphylaxis Patients (Experimental): Human amniotic mesenchymal stem cells (hAMSCs)
  Interventions: Other: Human amniotic mesenchymal stem cells

INTERVENTIONS:
Other: Human amniotic mesenchymal stem cells — 1. Intravenous infusion of hAMSCs: once every 3 weeks, a total of 6 times (if cured before the end of the planned course of treatment, it will be terminated in advance).
  2. Injection of hAMSCs to local skin lesions: once every 3 weeks, a total of 6 times (if cured before the end of the planned course of treatment, it will be terminated in advance).

SUMMARY:
Treatment for Uremic Calciphylaxis Patients with Human Amniotic Mesenchymal Stem Cells

DETAILED DESCRIPTION:
Calciphylaxis is a rare, devastating disorder causing excruciatingly painful ischemic skin lesions. Sepsis due to the infection of ulcerated wounds is a common cause of death. To date, practical therapies typically include wound care, pain management, anti-infection and aggressive treatment of predisposing conditions. Drugs such as sodium thiosulfate, bisphosphonate, and cinacalcet are also suggested. However, it's still a lethal disease with 1-year mortality up to 80% for dialysis patients. Here the investigators plan to treat uremic calciphylaxis patients with human amniotic mesenchymal stem cells (hAMSCs).

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old.
2. Patients with chronic kidney disease who did not or had regular dialysis (hemodialysis or peritoneal dialysis).
3. Clinical diagnosis of calciphylaxis.
4. All subjects signed informed consent.

Exclusion criteria:

1. Patients who refuse to sign informed consent.
2. Patients with malignant tumor or serious mental disease, cardiovascular disease, shock, abnormal liver function and secondary kidney disease.
3. Pregnant or lactating women of childbearing age.
4. Participation in another clinical trial with an experimental drug within 90 days prior the inclusion.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2022-09-17 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | Up to 1 year.
  The Bates-Jensen Wound Assessment (BWAT) is a standardized tool for quantitative assessment of wound healing that includes the 13 items listed below: (1)Size; (2)Depth; (3)Edges; (4)Undermining or pockets; (5)Necrotic tissue type; (6)Necrotic tissue amount; (7)Exudate type; (8)Exudate amount; (9)Surrounding skin color; (10)Peripheral tissue edema; (11)Peripheral tissue induration; (12)Granulation tissue; (13)Epithelialization.
  Each item was rated on a scale of 1 (best) to 5 (worst). The BWAT total score is the sum of the individual items with a possible range of 13 (best) to 65 (worst).

SECONDARY OUTCOMES:
Wound Pain | Up to 1 year.
  Assessed by pain visual analog scale (VAS). VAS Score is a horizontal line, 100 mm in length, anchored by word descriptors at each end. The subject marked the point on the line that represented his/her perception of his/her current pain status. VAS Score was determined by measuring in millimeters from the left hand end of the line (no pain) to the point that the subject marked. VAS Score range 0 (best) to 100 (Worst).
Measured Quality of Life | Up to 1 year.
  The wound-quality of life(QoL) questionnaire measures the disease-specific, health related QoL of patients with chronic wounds. It consists of 17 items on impairments that are assessed in retrospect to the preceding 7 days and rated on a 0 (best) to 4 (worse) scale with possible responses from "not at all" to "very much". The total score is the average of the 17 responses.
Systemic Infection | Up to 1 year.
  Assessed by serum hypersensitive C-reactive protein level(hCRP, mg/L). Increased serum hCRP levels above normal ranges indicate infection.
Survival State | From date of treatment until the date of die, assessed up to 1 year.
  Survival time from the hAMSCs treatment started(momths)

CONTACTS AND LOCATIONS:
Overall Officials: Ningning Wang, Professor, Principal Investigator — The First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital; Jiayin Liu, Professor, Study Director — The First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital; Lianju Qin, Principal Investigator — The First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nigwekar SU, Thadhani R, Brandenburg VM. Calciphylaxis. N Engl J Med. 2018 May 3;378(18):1704-1714. doi: 10.1056/NEJMra1505292. No abstract available. PMID 29719190
- [Background] Seethapathy H, Brandenburg VM, Sinha S, El-Azhary RA, Nigwekar SU. Review: update on the management of calciphylaxis. QJM. 2019 Jan 1;112(1):29-34. doi: 10.1093/qjmed/hcy234. PMID 30304522
- [Background] McCarthy JT, El-Azhary RA, Patzelt MT, Weaver AL, Albright RC, Bridges AD, Claus PL, Davis MD, Dillon JJ, El-Zoghby ZM, Hickson LJ, Kumar R, McBane RD, McCarthy-Fruin KA, McEvoy MT, Pittelkow MR, Wetter DA, Williams AW. Survival, Risk Factors, and Effect of Treatment in 101 Patients With Calciphylaxis. Mayo Clin Proc. 2016 Oct;91(10):1384-1394. doi: 10.1016/j.mayocp.2016.06.025. PMID 27712637
- [Background] Baby D, Upadhyay M, Joseph MD, Asopa SJ, Choudhury BK, Rajguru JP, Gupta S. Calciphylaxis and its diagnosis: A review. J Family Med Prim Care. 2019 Sep 30;8(9):2763-2767. doi: 10.4103/jfmpc.jfmpc_588_19. eCollection 2019 Sep. PMID 31681640
- [Background] Peng T, Zhuo L, Wang Y, Jun M, Li G, Wang L, Hong D. Systematic review of sodium thiosulfate in treating calciphylaxis in chronic kidney disease patients. Nephrology (Carlton). 2018 Jul;23(7):669-675. doi: 10.1111/nep.13081. PMID 28603903
- [Background] Udomkarnjananun S, Kongnatthasate K, Praditpornsilpa K, Eiam-Ong S, Jaber BL, Susantitaphong P. Treatment of Calciphylaxis in CKD: A Systematic Review and Meta-analysis. Kidney Int Rep. 2018 Oct 9;4(2):231-244. doi: 10.1016/j.ekir.2018.10.002. eCollection 2019 Feb. PMID 30775620
- [Background] Torregrosa JV, Sanchez-Escuredo A, Barros X, Blasco M, Campistol JM. Clinical management of calcific uremic arteriolopathy before and after therapeutic inclusion of bisphosphonates. Clin Nephrol. 2015 Apr;83(4):231-4. doi: 10.5414/CN107923. PMID 24075020
- [Derived] Naeem A, Gupta N, Naeem U, Khan MJ, Elrayess MA, Cui W, Albanese C. A comparison of isolation and culture protocols for human amniotic mesenchymal stem cells. Cell Cycle. 2022 Aug;21(15):1543-1556. doi: 10.1080/15384101.2022.2060641. Epub 2022 Apr 12. PMID 35412950
- See also: Related Info — http://www.nejm.org/doi/full/10.1056/NEJMra1505292
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/30304522
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/27712637
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/31681640
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/28603903
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/30775620
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/24075020/